CLINICAL TRIAL: NCT04277000
Title: Assessment of the Fall Risk Profile and Quality of Life of Subjects Aged 65 or Older Visiting the French Balaruc-les-bains Climatic Health Resort
Brief Title: Determinants of the Fall Risk Profile and Quality of Life of Older Subjects Visting Climatic Health Resorts
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL16_0129
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Fall; Fatigue
Keywords: Injurious falls; Fear of falling; Quality of life; Physical activity
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the study conducted in subjects aged 65 or older visiting the French Balaruc-les-bains climatic health resort was to :

* Determine factors that distinguish fallers from not fallers
* Determine factors that may predict falls and injurious falls, 3 and 6 months after the stay in the resort
* Determine the effects of the 3-week stay in the health resort on quality of life, fear of falling, fatigue, and physical activity

DETAILED DESCRIPTION:
In all subjects aged 65 or older visiting consecutively the resort over a 5-month period, a questionnaire was administered in order to record:

* The number of falls and injurious falls in the previous 12 months. Injurious falls are falls complicated by serious or moderate injuries. Falls with serious injuries were those that caused fractures, head injuries requiring admission to hospital, joint dislocations, sprains accompanied by reduced physical function, other non-specified serious joint injuries, and lacerations requiring sutures. Falls with moderate injuries were those that resulted in bruising, sprains, cuts, abrasions, or reduction in physical function for at least three days or in medical help
* Physical activity over the last 7 days, using the International Physical Activity Questionnaires (IPAQ)
* Fear of falling, using a visual analogue scale (VAS) (0 to 10).
* The feeling of fatigue over the previous month, using a visual analogue scale (0 to 10) A questionnaire was administered to record quality of life (EQ-5D-3L), at baseline and 7 days after the end of the stay A questionnaire snt by mail was filled in by subjects 3 and 6 months after the stay in the resort in order to record falls and injurious falls, fatigue, fear of falling, and physical activity (using the above questionnaires).

Physical measurements were performed at the entrance of the health resort :

* Body height and body weight to the nearest 0.5 cm and 0.1 kg to calculate the body mass index (kg.m-2)
* The Timed Up and Go test and the time to walk 4 meters at usual pace (Lusardi-2017)
* The 5 repeated chair stand test
* The maximum grip strength: using a Camry Electronic Hand Dynamometer
* The one-leg stand test (lowest value on the right and the left leg), and stand tests feet together, in semi-tandem, and tandem position
* The score of the Short Physical Performance Battery (SPPB) was calculated based on results of the 4-meter gait speed, and the 5-chair stand and balance tests
* The Fried's frailty phenotype score was calculated, based on - the weight loss in prior year (body weight at baseline ˗ the self-assessed body weight 12 months before inclusion) (1 point if ≥ 10 lbs lost unintentionally); - muscle strength (1 point if the maximum grip strength was low based on the dynamometer manual); - self-reported fatigue (1 point if Visual Analog Fatigue Scale ≥ 5 in men and ≥ 4 in women), - walking speed (1 point if 4-m walking speed at comfortable pace was in the lowest quintile of values of subjects with the same gender) (≤ 0.71 m.s-1 in women and ≤ 0.76 m.s-1 in men), - physical activities in the previous week (1 point if in the lowest quintile of values of IPAQ of subjects with the same gender) (≤ 2076 MET (Metabolic Equivalent Task) in women and ≤ 2320 MET in men). A total score of ≥ 3 points was indicative of frailty, 1 or 2 points of prefrail phenotype and a score of 0 is indicative of robustness

ELIGIBILITY:
Inclusion criteria:

* Patients aged 65 years or older visiting the Balaruc-les-bains resort for venous or rheumatologic complaints over the 5-month recruitment period
* Subjects able to comply with all trial procedures
* Subjects covered by public health insurance
* Signed informed

Exclusion criteria:

* Patients with severe physical or neuropsychiatric impairment making impossible the physical measurements at baseline or the reply to the questionnaires at baseline and during the 7 days-, 3 month-, and 6-month follow-up after the stay in the health resort.
* Subject unable to read or/and write

  * Subject who are in a dependency or employment with the sponsor or the investigator
  * Participation in another clinical trial within the last 4 weeks before the screening date

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects (women or men) aged 65 or older who consecutively visited the Balaruc-les-bains health resort for venous or rheumatologic complaints over a 5-month period
Sampling Method: Non-Probability Sample
Enrollment: 1471 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of new falls over the folly-up period | 1 year
  A fall is defined as an "unexpected event in which the participant comes to rest on the ground, floor, or other lower level" (J Am Geriatr Soc 2011;59:148-57)

SECONDARY OUTCOMES:
Number of injurious falls over the folly-up period | at 7 days, 3, and 6 months after the stay in the resort
  Number of injurious falls over the folly-up period (El Khoury F, 2015)
Fear of falling using a visual analogue scale | at 7 days, 3, and 6 months after the stay in the resort
  Fear of falling using a visual analogue scale (VAS) (0 to 10)(Scheffer-2010).
Feeling of fatigue using a visual analogue scale | at 7 days, 3, and 6 months after the stay in the resort
  the feeling of fatigue using a visual analogue scale (0 to 10)(Wolfe-2004; Hewlett-2011)

CONTACTS AND LOCATIONS:
Overall Officials: hubert Blain, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC